CLINICAL TRIAL: NCT02531581
Title: Comparing a Diuretic Vascular Filling in the Initial Management of Acute Pulmonary Embolism With Right Ventricular Dysfunction Normotensive
Brief Title: Diuretic Vascular Filling in the Initial Management of Acute PE With Right Ventricular Dysfunction Normotensive
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14-AOI-11
Record Dates: First submitted 2015-02-20; First posted 2015-08-24 (Estimated); Last update posted 2020-09-25 (Actual); Status verified 2018-02

CONDITIONS: Pulmonary Embolism
MeSH Terms: conditions — Pulmonary Embolism | interventions — Furosemide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Furosémide (Experimental): Furosemide: a dose of 40 mg IV bolus initially and live according to the diuretic response: possibility of 2nd Live IV bolus 40 mg if urine output <500 cc / 24 at the 4th hour.
  Establishment of an infusion G5 500cc% in "vein custody."
  Interventions: Drug: Furosemide
- NaCl 9% isotonic (Active Comparator): Infusion of 500 cc of isotonic NaCl 9% in 4 hours and 1000 cc 24-hour peripheral vein. The filling is being used in an "empirical" in severe EP and this group is therefore the control group.
  Interventions: Drug: NaCl 9% isotonic

INTERVENTIONS:
Drug: Furosemide — furosemide 40 mg bolus with second bolus to 4 hours so inadequate diuretic response defined as urine output <500cc
  Other Names: diuretic vascular filling
  Arms: Furosémide
Drug: NaCl 9% isotonic — normal saline 500 cc / 4 hours and 1 L / 24 hours
  Other Names: fluid replacement
  Arms: NaCl 9% isotonic

SUMMARY:
Pulmonary embolism (PE) is a serious disease with frequent intra hospital mortality remains high. If anticoagulation is perfectly codified, the remainder of the initial management has been less studied.

In particular, the "conditioning" Initial often involves systematic plasma volume of 250 to 500 cc, by analogy to other situations. But this treatment option is not based on factual data. In the right ventricular dysfunction that often accompany severe EP, volume expansion may instead be harmful, according to the law of Frank Starling. A retrospective study has recently shown a benefit of diuretic therapy in patients hospitalized for severe normotensive EP.

The proposed study is interventional, prospective, multicenter, randomized, require to include 60 patients.

The main objective of the study is the comparison of the troponin normalization period Ic (biomarker of right ventricular dysfunction) in patients hospitalized in the initial phase of a serious normotensive EP, between the 2 groups diuretic and filling Vascular.

The primary endpoint is the time in hours standardization of troponin Ic.

The secondary endpoints will be:

* the period of normalization of Brain Natriuretic Peptide (BNP)
* changes in echocardiographic parameters of right ventricular dysfunction
* a composite endpoint: cardiovascular death / cardiogenic shock / use of amines / use of thrombolysis.

DETAILED DESCRIPTION:
Main objective:

Compared with the time of normalization of cTnI (biomarker of right ventricular dysfunction) in hospitalized patients in the initial phase of a serious EP normotensive between the 2 groups diuretic and vascular filling

PRINCIPAL INCLUSION CRITERIA

* older than 18 Patient
* Hospitalized in the first 24 hours of a serious EP normotensive formally diagnosed (by a chest CT)

The serious nature without hypotension is defined by the presence of:

* From biological criteria: troponin and / or BNP positive AND
* In sonographic criteria: dilated right ventricle defined by echocardiography right over left ventricle ratio (VG)> 0.9 in apical 4- chamber or 0.7 in large parasternal axis and right ventricular systolic dysfunction (TAPSE <16 mm and S 'pulsed TDI tricuspid <10 cm / sec) or pulmonary arterial hypertension (PAH) Pulmonary Arterial Pressure with systolic (PAPs)> 35 mmHg or paradoxical septum

  * Informed consent signed
  * Affiliation to social security

PRINCIPAL EXCLUSION CRITERIA

* Thrombolysis before inclusion
* State of cardiogenic shock defined as systolic BP <90 mmHg or a drop of> 40 mmHg in systolic BP for> 15 minutes
* severe chronic renal impairment defined by clearance <30 ml / min.
* pregnant or nursing woman (a pregnancy test will be performed for XML File Identifier: cthC5Fc14NkHBXHkFCiTvGcJ8a8= Page 15/26 women of childbearing age and the results will be communicated to the patient by a doctor of his choice)
* Most People under guardianship
* hospitalized without their consent and not protected by law No
* Private person of liberty
* Residence time of more than 24 hours in another department after the positive diagnosis of pulmonary embolism

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized in the first 24 hours of a serious EP normotensive formally diagnosed (by a chest CT)

The serious nature without hypotension is defined by the presence of:

* From biological criteria: troponin and / or BNP positive AND
* In sonographic criteria: dilated right ventricle defined by echocardiography right over left ventricle ratio (VG)> 0.9 in apical 4- chamber or 0.7 in large parasternal axis and right ventricular systolic dysfunction (TAPSE <16 mm and S 'pulsed TDI tricuspid <10 cm / sec) or pulmonary arterial hypertension (PAH) Pulmonary Arterial Pressure with systolic (PAPs)> 35 mmHg or paradoxical septum
* Informed consent signed
* Affiliation to social security

Exclusion Criteria:

* Thrombolysis before inclusion
* State of cardiogenic shock defined as systolic BP <90 mmHg or a drop of> 40 mmHg in systolic BP for> 15 minutes
* severe chronic renal impairment defined by clearance <30 ml / min.
* pregnant or nursing woman (a pregnancy test will be performed for XML File Identifier: cthC5Fc14NkHBXHkFCiTvGcJ8a8=
* women of childbearing age and the results will be communicated to the patient by a doctor of his choice)
* Most People under guardianship
* hospitalized without their consent and not protected by law No
* Private person of liberty
* Residence time of more than 24 hours in another

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-12-23 (Actual); Primary Completion 2020-04-09 (Actual); Study Completion 2020-04-09 (Actual)

PRIMARY OUTCOMES:
Time normalization hours Troponin Ic. | participants will be followed for the duration of hospital stay, an expected average of 12 hours
  This is a direct assay on peripheral venous sampling, easy to collect, accurate and reproducible, made routines in biochemistry laboratories CHU Nice and Antibes CH. Assay kits are the same at the University Hospital of Nice and Antibes CH (BECKMANTM kit). The threshold of positivity of troponin is 0.07 ng / mL.

CONTACTS AND LOCATIONS:
Overall Officials: Emile FERRARI, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (1):
- CHU de Nice, Nice, France

REFERENCES:
- [Derived] Ferrari E, Sartre B, Labbaoui M, Heme N, Asarisi F, Redjimi N, Fourrier E, Squara F, Bun S, Berkane N, Breittmayer JP, Doyen D, Moceri P. Diuretics Versus Volume Expansion in the Initial Management of Acute Intermediate High-Risk Pulmonary Embolism. Lung. 2022 Apr;200(2):179-185. doi: 10.1007/s00408-022-00530-5. Epub 2022 Apr 5. PMID 35381867